CLINICAL TRIAL: NCT03813355
Title: Evaluation of tDCS Efficacy in Enduring Anorexia Nervosa : a Randomized Controlled Clinical Trial
Brief Title: Evaluation of tDCS Efficacy in Enduring Anorexia Nervosa
Acronym: EVASTRAM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of inclusion to meet the evaluation criteria
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1708195; 2018-A02866-49 (Other: ANSM)
Record Dates: First submitted 2018-12-20; First posted 2019-01-23 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-02

CONDITIONS: Anorexia Nervosa
Keywords: brain stimulation; Body Mass Index
MeSH Terms: conditions — Anorexia Nervosa | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active stimulation (Experimental): Brain stimulation by Transcranial Direct Current Stimulation (tDCS) with active stimulations
  Interventions: Device: transcranial Direct Current Stimulation (tDCS)
- Sham stimulation (Sham Comparator): Brain stimulation by Transcranial Direct Current Stimulation (tDCS) with inactive stimulations
  Interventions: Device: transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: transcranial Direct Current Stimulation (tDCS) — transcranial Direct Current Stimulation (tDCS) during 20 sessions

SUMMARY:
Approximately 20% of anorexia nervosa cases do not respond to conventional management strategies: cognitive behavioral therapy, weight gain contract, drug treatments, etc ... - whether they are applied outpatients or during very long hospitalizations. These situations of chronic evolution are characterized by a high rate of mortality. Brain stimulation could be an alternative therapy for these patients. tDCS (transcranial direct current stimulation) is a non-invasive stimulation technique that has demonstrated beneficial effects in other psychiatric conditions such as major depression or schizophrenia.

The objectives of the study will be to evaluate the efficacy of tDCS in anorexia nervosa resistant to conventional treatments on weight gain, eating behavior, psychological and nutritional behavioral scales, cognition, connectivity and brain activity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 anorexia nervosa criteria
* Body Mass Index (BMI) < 17kg/m2
* Conventional treatment failure over the last 12 months
* Refusal or no indication of artificial nutrition

Exclusion Criteria:

* Artificial nutrition
* Other chronic diseases
* drug use (except tobacco)
* pregnancy
* Edinburgh score < 14

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | weeks 8
  Change in body mass index after stimulation sessions. Weight and Height will be combined to report BMI in kg/m^2

SECONDARY OUTCOMES:
Eating Disorder Inventory (EDI) | weeks 8
  Change in Eating Disorder Inventory scale after stimulation sessions
  EDI measures :
  * Drive for thinness (score between 0-4)
  * Bulimia (score between 0-5)
  * Body dissatisfaction (score between 3-10)
  * ineffectiveness (score between 0-6)
  * Perfectionism (score between 0-5)
  * Interpersonal Distrust (score between 0-6)
  * Interoceptive awareness (score between 0-4)
  * Maturity Fears (score between 0-6)
Dutch Eating Behavior Questionnaire (DEBQ) | weeks 8
  Change in Dutch Eating Behavior Questionnaire (DEBQ) after stimulation sessions
  DEBQ measures :
  * Restrained eating (score between 10-30)
  * Emotional eating (score between 17-35)
  * external eating (score between 20-40)
Beck Depression Inventory (BDI) | weeks 8
  Change in Beck Depression Inventory after stimulation sessions.
  BDI measures :
  * No depression : score between 0-9
  * midl depression or anxiety : score between 10-19
  * moderate depression or anxiety : score between 20-25
  * moderate to severe depression or anxiety : score between 26-29
  * severe depression or anxiety : score between 30-40
  * very severe depression or anxiety : score between 41-84
State-Trait Anxiety Inventory (STAI) | weeks 8
  Change in State-Trait Anxiety Inventory (STAI) after stimulation sessions
  STAI measures :
  * no anxiety : score between 0-19
  * very low anxiety : score between 36-45
  * low anxiety : score between 46-55
  * moderate anxiety : score between 56-65
  * high anxiety : score between 56-65
  * very high anxiety : score greater than 65

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Massoubre, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (4):
- France (4):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - Hospices Civils de Lyon, Lyon
  - CHU Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No